CLINICAL TRIAL: NCT02845531
Title: Implantable Cardioverter Defibrillator Versus Optimal Medical Therapy In Patients With Variant Angina Manifesting as Aborted Sudden Cardiac Death
Acronym: VARIANT ICD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kee-joon Choi (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Kee-joon Choi, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-15
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Angina Pectoris, Variant; Sudden Cardiac Death
Keywords: Variant angina; Aborted sudden cardiac death; Implantable Cardioverter Defibrillator; Optimal Medical Therapy; ICD
MeSH Terms: conditions — Angina Pectoris, Variant; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICD implantation and optimal medical therapy (Experimental)
  Interventions: Device: Implantable Cardioverter Defibrillator
- optimal medical therapy (Active Comparator)
  Interventions: Drug: Optimal Medical Therapy

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator — Implantable Cardioverter Defibrillator and Optimal Medical Therapy
  Arms: ICD implantation and optimal medical therapy
Drug: Optimal Medical Therapy
  Arms: optimal medical therapy

SUMMARY:
The purpose of this study is to determine whether ICD(Implantable Cardioverter Defibrillator) implantation on the top of optimal medical therapy in patients with variant angina manifesting as aborted sudden cardiac death reduces the incidence of the death from any cause compared with optimal medical therapy alone.

DETAILED DESCRIPTION:
All participants will be monitored over a span of five years and the time point of the year of last subject last visit. The term "year of last subject last visit" refers to the time point of the last visit for all participants. At this specific time point, event occurrence check will be conducted to determine the occurrence of endpoint events among all participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients experienced successfully resuscitated cardiac arrest due to documented ventricular fibrillation or sustained rapid ventricular tachycardia
* Diagnosed as variant angina, defined by spontaneous coronary spasm with ST elevation (≥0.1mV) in the coronary angiogram and/or documented coronary spasm on ergonovine provocation coronary angiography

Exclusion Criteria:

* Significant (>50%) coronary artery stenosis on coronary angiography
* Organic heart disease known to be associated with sudden cardiac arrest.

  * Heart failure with reduced ejection fraction (Left Ventricular Ejection Fraction < 35%)
  * Presence of LV akinesia or aneurysm
  * Hypertrophic cardiomyopathy
  * Arrhythmogenic right ventricular dysplasia
* Chronic Heart Failure New York Heart Association functional class III or IV
* prior history of atrial or ventricular arrhythmia requiring class I or III antiarrhythmic drugs (flecainide, propafenone, amiodarone, sotalol and dronedarone)
* Prior catheter ablation for ventricular arrhythmia
* Primary cardiac electrical diseases (long QT syndrome, Brugada syndrome, catecholaminergic polymorphic ventricular tachycardia)
* Prior pacemaker or Implantable Cardioverter Defibrillator
* 2nd or 3rd degree AV block not related to coronary ischemia, requiring permanent pacemaker
* Patients with poor neurologic outcome (defined as cerebral performance category scale ≥3)
* Life expectancy <2 years
* Psychiatric illnesses that may be aggravated by device implantation or that may preclude systematic follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-11-29 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | 5 years

SECONDARY OUTCOMES:
Event rate of Cardiac death | 5 years
Event rate of Death from arrhythmia | 5 years
Event rate of Cardiac arrest | 5 years
Event rate of Recurrence of ventricular tachyarrhythmia | 5 years
Event rate of Hospitalization | 5 years
  Hospitalization due to unstable angina, acute myocardial infarction, heart failure, cardiac arrhythmia
Event rate of Appropriate ICD therapies | 5 years
  Appropriate ICD therapies defined as device-administered antitachycardia or defibrillation treatment for ventricular tachyarrhythmia that had not terminated spontaneously
Event rate of Inappropriate ICD therapies | 5 years
Event rate of Major device-related complications | 5 years
Event rate of Stroke | 5 years

CONTACTS AND LOCATIONS:
Locations (25):
- South Korea (25):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Busan National University Yangsan Hospital, Busan
  - Busan University Hospital, Busan
  - Dong-A Medical Center, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Chungnam National University Sejong Hospital, Sejong
  - Seoul university Bundang hospital, Seongnam
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Kangdong KyungHee University hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic Univ. of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided